CLINICAL TRIAL: NCT06948305
Title: Exploring the Care Needs of Spouses of Gynecological Cancer Patients and Evaluating the Development of Care Plans
Brief Title: Evaluate the Effectiveness of the Mobile Instant Messaging Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Hung-Ru Lin, PhD, RN, Distinguished Professor & Dean, College of Nursing, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NTUNHS-2025-04
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Gynecological Cancer

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- instant messaging software (Experimental)
  Interventions: Behavioral: instant messaging software
- "Control Group" (No Intervention)

INTERVENTIONS:
Behavioral: instant messaging software — instant messaging software
  Arms: instant messaging software

SUMMARY:
This study explores the caregiving needs of male spouses and develops an instant messaging software intervention to provide effective support. The goal is to help male spouses better adjust to their caregiving roles, reduce psychological stress and emotional distress, and improve overall health.

A randomized controlled trial will be conducted to evaluate the effectiveness of the mobile instant messaging intervention, analyzing its impact on reducing psychological distress and improving the quality of life of male spouses.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older, with a diagnosis of gynecological cancer (including cancers of the cervix, endometrium, fallopian tubes, ovaries, uterus, or vagina), and whose spouse has not been diagnosed with any other type of cancer;
2. The spouse has undergone cancer treatment, including surgery, chemotherapy, or radiotherapy;
3. Clear consciousness and ability to communicate in Mandarin or Taiwanese;
4. Willingness to participate in the study after being informed of the study purpose and procedures.

Exclusion Criteria:

Individuals with psychiatric disorders.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Supportive Care Needs -Partners & Caregivers 45, SCNS-P&C45 | Post-intervention assessments will be conducted at 1 month, 3 months, and 6 months after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Shin Kong Memorial Wu Ho-Su Hospital, Taipei, Taiwan